CLINICAL TRIAL: NCT03221400
Title: A Phase 1/2a, Open-label, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Anti-tumor Activity of PEN-866 in Patients With Advanced Solid Malignancies
Brief Title: PEN-866 in Patients With Advanced Solid Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tarveda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEN-866-001
Record Dates: First submitted 2017-07-13; First posted 2017-07-18 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Carcinoma; Endometrial Adenocarcinoma; Neoplasms; Squamous Cell Carcinoma of the Anus; Adenocarcinoma of the Pancreas; Advanced Cancer; Solid Tumor; Solid Carcinoma; Squamous Cell Carcinoma of the Cervix; Squamous Cell Carcinoma; Squamous Cell Carcinoma of the Vulva; Squamous Cell Carcinoma of the Penis; Gastric Cancer; Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Small-cell Lung Cancer; Small Cell Lung Carcinoma; Pancreatic Ductal Adenocarcinoma; Pancreatic Adenocarcinoma
MeSH Terms: conditions — Carcinoma; Neoplasms; Anus Neoplasms; Carcinoma, Squamous Cell; Stomach Neoplasms; Small Cell Lung Carcinoma | interventions — Fluorouracil; Leucovorin; niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1a PEN-866 Sodium (Single Agent) (Experimental): Dose escalation of PEN-866 Sodium administered intravenously
  Interventions: Drug: PEN-866 Sodium
- Phase 1b PEN-866 Sodium + Flurouracil + Folinic Acid (Experimental): Dose escalation of intravenous administration of PEN-866 Sodium in combination with fluorouracil and folinic acid
  Interventions: Drug: PEN-866 Sodium; Drug: fluorouracil; Drug: Folinic acid
- Phase 2a PEN-866 Sodium (Single Agent) (Experimental): Intravenously administered PEN-866 Sodium at the Recommended Phase 2 Dose
  Interventions: Drug: PEN-866 Sodium
- Phase 1b PEN-866 Sodium + Niraparib (Experimental): Dose escalation of intravenous administration of PEN-866 Sodium in combination with niraparib
  Interventions: Drug: PEN-866 Sodium; Drug: Niraparib

INTERVENTIONS:
Drug: PEN-866 Sodium — PEN-866 Sodium is a miniaturized conjugate that comprises an HSP90 targeting ligand linked to SN-38, the active metabolite of irinotecan. PEN-866 is available as a sterile lyophilized powder for solution for infusion.
Drug: fluorouracil — Fluorouracil 2400 mg/m2 IV
  Other Names: 5-Fluorouracil; 5-FU
  Arms: Phase 1b PEN-866 Sodium + Flurouracil + Folinic Acid
Drug: Folinic acid — Folinic acid 400 mg/m2 IV
  Other Names: Leucovorin
  Arms: Phase 1b PEN-866 Sodium + Flurouracil + Folinic Acid
Drug: Niraparib — Niraparib
  Other Names: Zejula
  Arms: Phase 1b PEN-866 Sodium + Niraparib

SUMMARY:
Protocol PEN-866-001 is an open-label, multi-center, first-in-human Phase 1/2a study evaluating PEN-866 in patients with advanced solid malignancies whose disease has progressed after treatment with previous anticancer therapies.

DETAILED DESCRIPTION:
Phase 1a will employ an adaptive model guided with overdose control principle to make dose recommendations and estimate the maximum tolerated dose (MTD) of PEN-866 (single agent).

Phase 1b will employ a standard 3 + 3 design to make dose recommendations and estimate the MTD of PEN-866 in combination therapy.

Phase 2a (single agent) will assess the safety, tolerability, pharmacokinetic, and pharmacodynamics profile of PEN-866 (single agent) at the recommended Phase 2 dose determined at the conclusion of Phase 1a in patients with advanced solid malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. M/F at least 18 years old
2. Performance status 0 or 1
3. Adequate bone marrow, liver, and kidney function within 28 days prior to first dose
4. Serum potassium, calcium, magnesium, phosphorus within normal limits
5. Adequate birth control
6. Central venous access line is required
7. Patients in Phase 1a must also have confirmed advanced solid malignancy that has progressed after one or more prior lines of anticancer therapy and no other standard of care therapies that are deemed appropriate for treatment of their malignancy
8. Patients in Phase 2a must have measurable disease per RECIST 1.1 and documented disease progression during or after their most recent line of anticancer therapy.
9. Patients in Phase 2a must have disease history specific to their disease as listed below:

   * Small Cell Lung Cancer (SCLC): Patients with locally recurrent or metastatic SCLC whose disease has progressed after having received one or more prior lines of chemotherapy.
   * Gastric or gastroesophageal (GEJ) adenocarcinoma: Patients with locally recurrent or metastatic gastric or GEJ adenocarcinoma whose disease has progressed after having received one or more prior lines of chemotherapy.
   * Squamous cell carcinoma (SCC) of the genitalia (anus, cervix, vulva, or penis): Patients with locally recurrent or metastatic SCC of the genitalia (anus, cervix, vulva, or penis) whose disease has progressed after having received one or more prior lines of chemotherapy, including those whose disease has progressed after postoperative adjuvant chemotherapy or neoadjuvant chemotherapy prior to radiation or surgery.
   * Pancreatic adenocarcinoma (PDAC): Patients with locally recurrent or metastatic PDAC whose disease has progressed after having received one or more prior lines of chemotherapy, including those whose disease has progressed within 6 months of postoperative adjuvant chemotherapy.
   * Endometrial adenocarcinoma (EC): Patients with locally recurrent or metastatic EC whose disease has progressed after having received one or more prior lines of chemotherapy, including those whose disease has progressed within 6 months of postoperative adjuvant chemotherapy.
10. For Phase 1b patients receiving PEN-866 in combination with fluorouracil and folinic acid only:

    * Patients with metastatic PDAC who have progressed after having received one or more prior lines of chemotherapy, including those whose disease has progressed within 6 months of postoperative adjuvant chemotherapy.
11. For Phase 1b patients receiving the Niraparib combination only:

    * Patients must have confirmed advanced solid malignancy that has progressed after one or more prior lines of anticancer therapy and no other standard of care therapies that are deemed appropriate for treatment of their malignancy

Exclusion Criteria:

1. Treatment with anticancer therapy or investigational drug or device within 2 wk (6 wk for nitrosureas or mitomycin C) before C1D1, and any drug-related toxicities must have recovered to grade 1 or less with the exception of alopecia and peripheral neuropathy.
2. Phase 2a only: Prior treatment with topoisomerase I inhibitor(s).
3. Cardiac disease such as unstable angina within 6 months of screening, myocardial infarction within 6 months of screening, NY Heart Association Class III - IV heart failure, QTc greater than 470 msec, congenital long Qt syndrome, symptomatic orthostatic hypotension within 6 months of screening, uncontrolled hypertension, or clinically important abnormalities in heart rhythm, conduction, morphology of resting ECG.

   -For Phase 1b patients receiving the Niraparib combination only: hypertension as defined as diastolic > 90 mmHg or systolic > 140 mmHg
4. Stroke or transient ischemic attack within 6 months of screening
5. Prior history of posterior reversible excephalopathy scyndrome (PRES).
6. Peripheral neuropathy greater than grade 2
7. Patients requiring medications with drugs that are inhibitors of UGT1A1 or substrates of CYP1A2, P-gP, BCRP, OATP1B1, OATP1B3 or OCT1 transporters
8. Leptomeningeal disease or spinal cord compression unless controlled and asymptomatic with surgery, radiation, and not requiring steroids within 4 weeks prior to C1D1.
9. Brain metastases unless previously treated and asymptomatic. Stable low dose of steroids is permitted.
10. Major surgery within 28 days of first drug dose
11. If female, pregnant or breast feeding
12. Evidence of severe uncontrolled systemic disease, bleeding diatheses, renal or liver transplant, active infection with hep B or C or HIV
13. Hypersensitivity or anaphylactic reaction to ganetespib or other HSP90 inhibitors, irinotecan, SN-38 or its derivatives
14. Any medical, psychological, or social condition that would interfere with the patient's participation in the study.
15. Live virus and bacterial vaccines administered within 30 days prior to C1D1.
16. Any medical, psychological, or social condition that would interfere with the patient's participation in the study.

    For Phase 1b patients receiving niraparib combination only, the following additional exclusion criteria apply:
17. Prior treatment with niraparib.
18. Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones, liver metastatses or otherwise stable chronic liver disease per investigator assessment).
19. Severe hepatic impairment.
20. Treatment with transfusions and/or erythropoietin for the treatment of anemia within 4 weeks prior to C1D1.
21. Any known or current diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
22. History of prostate cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2017-08-29 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1a and 1b : Incidence of Dose-Limiting Toxicities (DLTs) | Patients will be followed for 28 days to determine the incidence of DLTs.
  The Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) will be determined by assessing the incidence of DLTs and treatment related adverse events of PEN-866 as a single agent (Phase 1a) or in combination therapy (Phase 1b).
All Phases: Incidence of treatment related adverse events (Safety and tolerability) | From date of first treatment/trial entry up to 28 days following the last treatment.
  Safety and tolerability will be determined by assessing the incidence of treatment related adverse events.
Phase 2a: Efficacy of PEN-866 in patients with SCLC using best overall response rate | From the date of first treatment through the date of first documented progression, assessed up to (estimated) 18 months
  Efficacy of PEN-866 in patients with SCLC will be assessed using best overall tumor response rate defined as complete response (CR) or partial response (PR) according to RECIST 1.1.
Phase 2a: Efficacy of PEN-866 in patients with gastric or gastroesophageal junction (GEJ) adenocarcinoma using best overall response rate | From the date of first treatment through the date of first documented progression, assessed up to (estimated) 18 months
  Efficacy of PEN-866 in patients with gastric or GEJ adenocarcinoma will be assessed using best overall tumor response rate defined as CR or PR according to RECIST 1.1.
Phase 2a: Efficacy of PEN-866 in patients with pancreatic adenocarcinoma using Disease Control Rate (DCR) | From the date of first treatment through the date of first documented progression, assessed up to (estimated) 18 months
  Efficacy of PEN-866 in patients with pancreatic adenocarcinoma will be assessed using DCR defined as a best response of CR, PR, or stable disease (SD) according to RECIST 1.1.
Phase 2a: Efficacy of PEN-866 in patients with endometrial adenocarcinoma using best overall response rate | From the date of first treatment through the date of first documented progression, assessed up to (estimated) 18 months
  Efficacy of PEN-866 in patients with endometrial adenocarcinoma will be assessed using best over all tumor response rate defined as CR or PR according to RECIST 1.1.
Phase 2a: Efficacy of PEN-866 in patients with squamous cell carcinoma of the genitalia (anus, cervix, vulva, or penis) using best overall response rate | From the date of first treatment through the date of first documented progression, assessed up to (estimated) 18 months
  Efficacy of PEN-866 in patients with squamous cell carcinoma of the genitalia will be assessed using best over all tumor response rate defined as CR or PR according to RECIST 1.1.

SECONDARY OUTCOMES:
Maximum concentration (Cmax) of PEN-866 and its components (HSP90 ligand and SN-38) | 1 Month (Phase 1a); 14 days (Phase 1b); assessed up to (estimated) 18 months for Phase 2a
  Characterize the pharmacokinetic properties of PEN-866 and its components (HSP90 targeting ligand and SN-38)
Area under the curve (AUC) of PEN-866 and its components (HSP90 ligand and SN-38) | 1 Month (Phase 1a); 14 days (Phase 1b); assessed up to (estimated) 18 months for Phase 2a
  Characterize the pharmacokinetic properties of PEN-866 and its components (HSP90 targeting ligand and SN-38)
Half-life (t1/2) of PEN-866 and its components (HSP90 ligand and SN-38) | 1 Month (Phase 1a); 14 days (Phase 1b); assessed up to (estimated) 18 months for Phase 2a
  Characterize the pharmacokinetic properties of PEN-866 and its components (HSP90 targeting ligand and SN-38)
Phase 1b: Characterize the plasma pharmacokinetics (PK) of the combination therapies and their components | 14 days
  PK parameters (CMax, AUC) will be evaluated in plasma by standard non-compartmental methods (compartmental modeling may be performed if appropriate).
Phase 1a: Tumor response using RECIST 1.1 criteria | Baseline and every 6 weeks until date of first documented progression or death (estimated 6 months)
  Size of tumors by CT or MRI using tumor response criteria according to RECIST 1.1 and duration of response.
Phase 1b: Disease Control Rate | From date of first treatment through the date of date of first documented progression, assessed up to (estimated) 18 months
  Efficacy of PEN-866 in combination therapy will be assessed using DCR as defined as CR, PR, or SD according to RECIST 1.1.
Phase 2a: Disease Control Rate in patients with SCLC, gastric or gastroesophageal junction adenocarcinoma, endometrial adenocarcinoma, and squamous cell carcinoma of the genitalia (anus, cervix, vulva, and penis) | From date of first treatment through the date of date of first documented progression, assessed up to (estimated) 18 months
  Efficacy of PEN-866 in SCLC, gastric or gastroesophageal junction adenocarcinoma, endometrial adenocarcinoma, and squamous cell carcinoma of the genitalia (anus, cervix, vulva, and penis) will be assessed using DCR as defined as CR, PR, or SD according to RECIST 1.1.
Phase 2a: Evaluate the best overall response rate in patients with pancreatic adenocarcinoma | From date of first treatment through the date of first documented progression, assessed up to (estimated) 18 months
  Efficacy of PEN-866 in pancreatic adenocarcinoma using best overall tumor response rate as defined as CR or PR according to RECIST 1.1
Phase 1b and 2a: Duration of Response | From date of first treatment until the date of date of death from any cause, assessed up to (estimated) 18 months
  Time from first documented response (CR or PR) to date of first documented disease progression or death due to underlying cancer.
Phase 2a: Radiographic progression free survival | From date of first treatment until the date of first documented progression or date of death from any cause, whichever is first, assessed up to (estimated) 18 months
  Time from first PEN-866 dose to date of first documented progression or date of death from any cause, whichever came first
Phase 2a: Overall survival | From date of first treatment until the date of date of death from any cause, assessed up to (estimated) 18 months
  Time from first PEN-866 dose to date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Anish Thomas, MD, Study Chair — National Cancer Institute (NCI)
Locations (16):
- United States (16):
  - Highlands Oncology Group, Springdale, Arkansas
  - Sarah Cannon Reasearch Institute at HealthONE, Denver, Colorado
  - Florida Cancer Specialists - South, Fort Myers, Florida
  - Florida Cancer Specialists - North, St. Petersburg, Florida
  - Florida Cancer Specialists - East, West Palm Beach, Florida
  - National Institutes of Health / National Cancer Institute, Bethesda, Maryland
  - Henry Ford, Detroit, Michigan
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Stephenson Cancer Center, University of Oklahoma, Oklahoma City, Oklahoma
  - Sidney Kimmel Cancer Center at Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Prisma Health - Upstate, Greenville, South Carolina
  - The West Clinic, Germantown, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No